CLINICAL TRIAL: NCT01962571
Title: Treatment of Optic Neuritis With Erythropoietin: a Randomised, Double-blind, Placebo-controlled Trial
Acronym: TONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Eye Hospital, Freiburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Wolf Lagrèze, Prof. Dr. med., University Eye Hospital, Freiburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P000053; 2013-002515-10 (EudraCT Number); DRKS00005298 (Registry Identifier: German Clinical Trials Register (DRKS)); 01KG1306 (Other Grant/Funding Number: Federal Ministry of Education and Research)
Record Dates: First submitted 2013-09-30; First posted 2013-10-14 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Optic Neuritis
Keywords: Optic neuritis; Multiple Sclerosis; Clinically isolated syndrome; Erythropoietin
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin alfa (Experimental): Recombinant human EPO (Epoetin alfa HEXAL®) will be given as an i.v. bolus injection on days 1, 2 and 3. The dosage per day will be 33.000 IU in accordance with previous trials.
  Interventions: Drug: Erythropoietin alfa
- Placebo (Placebo Comparator): As matched placebo for this study, sterile normal saline (0.9% sodium chloride for i.v. administration) will be used. It will be given as a bolus injection in the same manner as EPO.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin alfa
  Arms: Erythropoietin alfa
Drug: Placebo
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This clinical trial aims at preventing visual dysfunction and optic nerve degeneration associated with autoimmune optic neuritis by systemic i.v. administration of 33.000 IU erythropoietin over 3 days. The primary objective is to determine the efficacy of erythropoietin compared to placebo given as add-on to methylprednisolone as assessed by measurements of retinal nerve fibre layer thickness and low contrast visual acuity 6 months after acute optic neuritis.

ELIGIBILITY:
Patients eligible for inclusion in this trial must meet all of the following criteria:

1. Written informed consent obtained according to international guidelines and local laws
2. Male and female patients aged ≥ 18 to ≤ 50 years
3. Patients with ON
4. First symptoms of ON ≤ 10 days prior to the first administration of investigational product
5. High contrast visual acuity (HCVA) of ≤ 0.5 (decimal system)
6. Adequate OCT measurements available

Patients eligible for this trial must not meet any of the following criteria:

1. Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial
2. Simultaneous participation in another interventional trial which could interfere with this trial and/or participation in a clinical trial within the last 3 months before enrolment in this trial
3. Refractive anomalies: Hyperopia > 5 dpt, myopia < -7 dpt, astigmatism > 3 dpt
4. Media opacity
5. Severe papillitis
6. Previous ON
7. Any other optic nerve and retinal disease
8. Pre-existing MS or any other neurological disease
9. Congenital diseases:

   * thrombophilia
   * phenylketonuria
10. Acquired diseases:

    * autoimmune diseases,
    * cardiovascular diseases,
    * diabetes mellitus,
    * uncontrolled hypertension (with blood pressure > 140 / 90 mm Hg (cf. chapter 7.7.5)),
    * any malignancy,
    * epilepsy,
    * known tuberculosis with ongoing or unknown activity,
    * acute gastrointestinal ulceration within the last 3 months prior to randomisation,
    * acute viral, bacterial or fungal infection,
    * known infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus, or Hepatitis C Virus,
    * history of colitis ulcerosa, diverticulitis, or acute enteroanastomosis,
    * known osteoporosis,
    * history of thromboembolic events,
    * elevated haemoglobin level (>17 g/dl in men or >15 g/dl in women)
    * polycythaemia
    * any other significant illness potentially interfering with any trial assessment or trial treatment
11. Performing semi-professional or professional sporting activities or physical training
12. Pre-treatment with corticosteroids in the last 30 days prior to the onset of optic neuritis
13. Pre-treatment with EPO
14. Known or persistent abuse of medication, drugs or alcohol
15. Active immunization within 2 weeks prior to randomisation
16. Significant surgery within 4 weeks prior to randomisation
17. Blood donation or bloodletting within 4 weeks prior to screening
18. Pre-treatment with immunosuppressive or immunomodulatory agents
19. Persons who are in a relationship of dependence/employment with the sponsor or the investigator

    This section concerns only female patients who are able to have a child:
20. Current or planned pregnancy; nursing period within 3 months from investigational product administration
21. Unwillingness to use one of the following safe combination methods of contraception within 3 months from investigational product administration to achieve a PEARL index of <1: female condom, diaphragm or coil, each used in combination with a spermicide; hormonal intra-uterine device or hormonal contraception in combination with a mechanical method of contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Global retinal nerve fibre layer thickness (RNFLT-G) | 6 months
  Determination of the efficacy of erythropoietin compared to placebo given as add-on to methylprednisolone (standard of care) as assessed by measurement of global retinal nerve fibre layer thickness (RNFLT-G) in the affected eye 6 months after randomisation.
Low contrast visual acuity (LCVA) | 6 months
  Determination of the efficacy of erythropoietin compared to placebo given as add-on to methylprednisolone (standard of care) as assessed by measurement of low contrast visual acuity (LCVA) in the affected eye 6 months after randomisation.

SECONDARY OUTCOMES:
Absolute values of the global retinal nerve fibre layer thickness | 6 months
Retinal nerve fibre layer thickness in the papillomacular bundle | 6 months
Retinal nerve fibre layer thickness in the temporal quadrant | 6 months
Total macular volume | 6 months
Visual acuity | 6 months
Contrast sensitivity | 6 months
Mean visual field defect | 6 months
Latency [ms] and amplitude [µV] of visual evoked potentials (VEP) | 6 months
Expanded Disability Status Scale (EDSS) score | 6 months
Quality of life | 6 months
  Determined by NEI-VFQ-25
Safety | Screening until end of study
  Assessment of AEs / SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Wolf A. Lagrèze, Prof., Principal Investigator — Eye Hospital, Medical Center - University of Freiburg
Locations (11):
- Germany (11):
  - Medical Center - University of Freiburg, Eye Hospital, Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg University Hospital, Department of Neurooncology, Heidelberg, Baden-Wurttemberg
  - Tuebingen University Hospital, Tübingen, Baden-Wurttemberg
  - University Hospital Erlangen, Erlangen, Bavaria
  - University Hospital of Munich, Munich, Bavaria
  - University Hospital Klinikum rechts der Isar, Munich, Munich, Bavaria
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - Hannover Medical School, Hanover, Lower Saxony
  - Duesseldorf University Hospital, Düsseldorf, North Rhine-Westphalia
  - University Medical Center of the Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate
  - University Medical Center Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Background] Suhs KW, Hein K, Sattler MB, Gorlitz A, Ciupka C, Scholz K, Kasmann-Kellner B, Papanagiotou P, Schaffler N, Restemeyer C, Bittersohl D, Hassenstein A, Seitz B, Reith W, Fassbender K, Hilgers R, Heesen C, Bahr M, Diem R. A randomized, double-blind, phase 2 study of erythropoietin in optic neuritis. Ann Neurol. 2012 Aug;72(2):199-210. doi: 10.1002/ana.23573. PMID 22926853
- [Background] Diem R, Molnar F, Beisse F, Gross N, Druschler K, Heinrich SP, Joachimsen L, Rauer S, Pielen A, Suhs KW, Linker RA, Huchzermeyer C, Albrecht P, Hassenstein A, Aktas O, Guthoff T, Tonagel F, Kernstock C, Hartmann K, Kumpfel T, Hein K, van Oterendorp C, Grotejohann B, Ihorst G, Maurer J, Muller M, Volkmann M, Wildemann B, Platten M, Wick W, Heesen C, Schiefer U, Wolf S, Lagreze WA. Treatment of optic neuritis with erythropoietin (TONE): a randomised, double-blind, placebo-controlled trial-study protocol. BMJ Open. 2016 Mar 1;6(3):e010956. doi: 10.1136/bmjopen-2015-010956. PMID 26932144
- [Derived] Kuchlin S, Ihorst G, Heinrich SP, Farassat N, Marquez Neila P, Hug MJ, Albrecht P, Lagreze WA. Clinical Predictors in Acute Optic Neuritis: Analysis Based on Clinical Trial Data. Ophthalmology. 2025 Jun;132(6):631-643. doi: 10.1016/j.ophtha.2025.01.010. Epub 2025 Jan 17. PMID 39827907
- [Derived] Kuchlin S, Ihorst G, Heinrich SP, Marquez Neila P, Albrecht P, Hug MJ, Diem R, Lagreze WA. Disease Course of Clinically Isolated Optic Neuritis. Neurol Neuroimmunol Neuroinflamm. 2024 May;11(3):e200223. doi: 10.1212/NXI.0000000000200223. Epub 2024 Apr 8. PMID 38588480
- [Derived] Kuchlin S, Ihorst G, Grotejohann B, Beisse F, Heinrich SP, Albrecht P, Ungewiss J, Worner M, Hug MJ, Wolf S, Diem R, Lagreze WA; TONE Study Group. Treatment With Erythropoietin for Patients With Optic Neuritis: Long-term Follow-up. Neurol Neuroimmunol Neuroinflamm. 2023 Apr 24;10(4):e200067. doi: 10.1212/NXI.0000000000200067. Print 2023 Jul. PMID 37094997
- [Derived] Lagreze WA, Kuchlin S, Ihorst G, Grotejohann B, Beisse F, Volkmann M, Heinrich SP, Albrecht P, Ungewiss J, Worner M, Hug MJ, Wolf S, Diem R; TONE study group. Safety and efficacy of erythropoietin for the treatment of patients with optic neuritis (TONE): a randomised, double-blind, multicentre, placebo-controlled study. Lancet Neurol. 2021 Dec;20(12):991-1000. doi: 10.1016/S1474-4422(21)00322-7. PMID 34800417
- [Derived] Wilhelm H, Schabet M. The Diagnosis and Treatment of Optic Neuritis. Dtsch Arztebl Int. 2015 Sep 11;112(37):616-25; quiz 626. doi: 10.3238/arztebl.2015.0616. PMID 26396053
- [Derived] Lagreze W, Diem R. [New aspects in the therapy of multiple sclerosis and optic neuritis]. Ophthalmologe. 2014 Aug;111(8):709-14. doi: 10.1007/s00347-013-2987-7. German. PMID 25063544